CLINICAL TRIAL: NCT03625544
Title: A Randomized Intra-Patient Controlled Trial of MagnetOs™ Granules vs. Autograft in Instrumented Posterolateral Spinal Fusion
Brief Title: MagnetOs™ Granules vs. Autograft in Instrumented Posterolateral Spinal Fusion
Acronym: MaxA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.C. Kruyt, MD, PhD (Other)
Collaborators: Kuros BioSciences B.V. (Industry)
Responsible Party: Sponsor-Investigator, M.C. Kruyt, MD, PhD, Orthopaedic surgeon, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL64652.041.18
Record Dates: First submitted 2018-07-02; First posted 2018-08-10 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Spinal Fusion
Keywords: bone graft; ceramic; spinal fusion; RCT

STUDY DESIGN:
Intervention Model Description: Intra-patient model, so each patient receives both conditions and serves as its own control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MagnetOs™ Granules (Experimental): MagnetOs™ Granules
  Interventions: Procedure: Instrumented posterolateral spinal fusion; Device: MagnetOs™ Granules
- Autograft (Active Comparator): Autologous bone graft
  Interventions: Procedure: Instrumented posterolateral spinal fusion; Procedure: Autologous bone graft

INTERVENTIONS:
Procedure: Instrumented posterolateral spinal fusion — Instrumented posterolateral spinal fusion, with or without an additional interbody device
Device: MagnetOs™ Granules — 8-10cc of MagnetOs™ Granules per spinal level at the randomized allocation side of the spine (left or right)
  Arms: MagnetOs™ Granules
Procedure: Autologous bone graft — 8-10cc autologous bone graft per spinal level at the control side of the spine (left or right). This can be a combination of local bone and iliac crest bone, but at least 50% of the volume has to be iliac crest bone graft.
  Arms: Autograft

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of MagnetOs™ Granules as an alternative to autologous bone graft in adult patients undergoing an instrumented posterolateral fusion of the thoracolumbar, lumbar or lumbosacral spine, in terms of efficacy and safety. After instrumentation and based on randomization, one side of the spine will be grafted with MagnetOs™ Granules and the other side with autologous bone graft. Thereby, each patient serves as its own control.

DETAILED DESCRIPTION:
Posterolateral spinal fusion is currently performed by using large amounts of autologous bone graft. Drawbacks of bone grafting include the need for an additional surgical procedure, limited supply, sub-optimal bone quality in osteoporotic patients and harvesting morbidity, which led to the development of numerous bone graft substitutes. Recently, a promising synthetic graft substitute has been developed that has shown favorable results in pre-clinical studies. This product, MagnetOs™ Granules, is CE-marked and received 510(k) clearance from the US Food and Drug Administration. The aim of the current study is to demonstrate non-inferiority of MagnetOs™ Granules compared to autograft in instrumented posterolateral spinal fusion, in terms of efficacy and safety.

This study is designed as a multicenter, observer blinded, randomized, controlled non-inferiority trial with intra-patient comparisons. A total of 100 adult patients qualified for posterolateral spinal fusion in the thoracolumbar and lumbosacral region (T10-S2) will be recruited and enrolled. According to a randomization scheme, one side of the spine will be grafted with the MagnetOs™ Granules and the other side with bone harvested from the iliac crest and local bone. The rest of the surgical procedure will be according to standard care.

The primary efficacy outcome is the rate of successful posterolateral spinal fusion after one year, assessed on CT-scans. Non-inferiority of the MagnetOs™ condition compared to the autograft condition will be assessed using a McNemar's test. The primary safety outcome is the number and nature of (serious) adverse events related to the surgical procedure compared to control populations from literature. Secondary outcomes are the comparison to its predicate (AttraX® Putty), relation between posterolateral fusion and interbody fusion after one-year, posterolateral spinal fusion rate after two years, relevance of iliac crest donor site pain and the incidence of long-term complication and relation with risk factors in the combined population of this study and a recently completed clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* To be treated with instrumented posterolateral thoracolumbar spinal fusion with the use of iliac crest bone, with or without additional posteriorly inserted interbody devices (PLIF, TLIF), because of (1) deformity, (2) structural instability and/or (3) expected instability as a result of decompression for spinal stenosis;

  1. Deformity is defined as a scoliosis in the coronal plane of >20° and/or a sagittal balance disturbance according the SRS/Schwab classification on standardized standing full spine radiographs;
  2. Preoperative instability is defined as a progressive angular deformity or spondylolisthesis in standing radiographs;
  3. Decompression for spinal stenosis is done in the occurrence of radiological evidence of stenosis on MRI and clinical leg and/or back pain with one or more of the following phenomena: radiculopathy, sensory deficit, motor weakness, reflex pathology or neurogenic claudication.
* Non-responsive to at least 6 months of non-operative treatment prior to study enrollment;
* Fusion indicated for one to six levels in the T10 to S2 region. In case of vertebral osteotomies (PSO or VCR) the osteotomized segment will not be included in the assessment of the fusion rate;
* Willing and able to understand and sign the study specific Patient Informed Consent;
* Skeletally mature between 18 and 80 years of age.

Exclusion Criteria:

* Any previous surgical attempt(s) for spinal fusion (revision surgery) of the intended segment(s);
* Previous treatments that compromise fusion surgery like irradiation;
* Previous autologous bone grafting procedures that compromise the quality and amount of iliac crest bone grafting;
* Indication for spinal fusion because of an acute traumatic reason, like a spinal fracture;
* Active spinal and/or systemic infection;
* Spinal metastasis in the area intended for fusion;
* Systemic disease or condition, which would affect the subjects ability to participate in the study requirements or the ability to evaluate the efficacy of the graft (e.g. active malignancy, neuropathy, pregnancy);
* At risk to be non-compliant e.g.: (recently treated for) substance abuse, detainee, likely to immigrate
* Participation in clinical trials evaluating investigational devices, pharmaceuticals or biologics within 3 months of enrollment in this study;
* Female patients who intend to be pregnant within 1.5 year of enrollment in the study;
* Body mass index (BMI) larger than 36 (morbidly obese);
* Being expected to require additional surgery to the same spinal region within the next 6 months;
* Current or recent (<1yr) corticosteroid use equivalent to prednisone ≥5mg/day, prescribed for more than 6 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Posterolateral spinal fusion rate at one-year follow-up | 1 year (12-15 months) after surgery
  For the efficacy analysis, a comparison will be made between the fusion performance of the MagnetOs™ Granules condition and the autograft condition after one year, assessed at CT-scans. Non-inferiority of MagnetOs™ Granules will be tested with a McNemar's test.
Rate of (serious) adverse events that are related to the spinal fusion procedure in any way, and their potential relation with MagnetOs™ Granules. | Until 2 years (22-26 months) after surgery
  The safety of MagnetOs™ Granules will be evaluated by comparing the number and nature of all (serious) adverse events that may in any way be related to the surgical procedure to rates in control populations from literature.

SECONDARY OUTCOMES:
Relation between successful posterolateral spinal fusion and interbody fusion at one-year follow-up | 1 year (12-15 months) after surgery
  Odds ratio for relation between posterolateral spinal fusion and interbody fusion assessed on CT-scans
Posterolateral spinal fusion rate at two years follow-up compared to the fusion rate at one-year follow-up | 2 years (22-26 months) after surgery
  Assessed on CT-scans
Posterolateral spinal fusion rate of MagnetOs™ Granules compared to the results of AttraX® Putty from a previous study (AxA study) | 1 year (12-15 months) after surgery
  Posterolateral spinal fusion rate of MagnetOs™ Granules vs. AttraX® Putty assessed on CT-scans
Relation between successful posterolateral spinal fusion and interbody fusion of MagnetOs™ Granules compared to the results of AttraX® Putty from a previous study (AxA study) | 1 year (12-15 months) after surgery
  Odds ratio for relation between posterolateral spinal fusion and interbody fusion of MagnetOs™ Granules vs. AttraX® Putty assessed on CT-scans
Effect of blinding on perceived donor site pain | Until 2 years (22-26 months) after surgery
  Visual analogue scale (VAS) scores for donor site pain reported by patients unblinded to the iliac crest donor site in comparison to these outcomes of the blinded patients from a previous study (AxA study)
Incidence of long-term complications and relation with risk factors in the combined population of this study and a previous study (AxA study) | Until 2 years (22-26 months) after surgery
  Like adjacent segment disease, in relation to length of construct and sagittal balance, and risk factors for failures

CONTACTS AND LOCATIONS:
Overall Officials: Moyo Kruyt, MD, PhD, Principal Investigator — UMC Utrecht
Locations (5):
- Netherlands (5):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - St. Antonius Hospital, Nieuwegein
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication of primary outcome — https://journals.lww.com/spinejournal/fulltext/2024/10010/efficacy_of_biphasic_calcium_phosphate_ceramic.1.aspx

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT03625544/Prot_SAP_000.pdf